CLINICAL TRIAL: NCT04644796
Title: A Randomized Controlled Trial of the Effect of Liposomal Bupivacaine (Exparel) When Compared to Saline Control in Reducing Opioid Utilization for Pain Management in Postoperative Lumbar Spine Surgeries.
Brief Title: A Randomized Trial of Exparel vs Saline in Opioid Reduction of Pain Management Following Lumbar Spine Surgeries.
Acronym: Exparel
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2037544
Record Dates: First submitted 2020-11-19; First posted 2020-11-25 (Actual); Results first posted 2023-01-04 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Lumbar Spine Degeneration
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned to either the treatment group or the placebo group. Patients in the study group will receive liposomal bupivacaine at the end of the procedure (following fascial closure, but prior to superficial closure), while patients in the placebo group will receive sterile saline. The injectate should be injected slowly and deeply, infusing ~1-2 mL according to manufacture guidelines for infiltration. According to these guidelines, injection should utilize a moving needle technique (inject while withdrawing the needle) at multiple locations surrounding the incision(s) to achieve maximal effect. Care will be taken to aspirate prior to injection to minimize the risk of intravascular injection of medication.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Liposomal bupivacaine can be differentiated visually from normal saline. In order to blind the surgeons from treatment vs control, the syringes containing the medication or saline will be sheathed by the investigational drug study department.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo Group (Placebo Comparator): Patients in this group will be given the placebo (sterile saline).
  Interventions: Drug: saline 0.9%
- Liposomal bupivacaine (Active Comparator): Patients in this group will be given the study drug (liposomal bupivacaine).
  Interventions: Drug: Liposomal bupivacaine

INTERVENTIONS:
Drug: saline 0.9% — Patients included in the placebo group will have their incisional site infused, targeting the paraspinal muscles with sterile saline at the end of their surgery.
  Other Names: sterile saline
  Arms: Placebo Group
Drug: Liposomal bupivacaine — Patients included in the treatment group will have their incisional site infused, targeting the paraspinal muscles with liposomal bupivacaine at the end of their surgery.
  Other Names: Exparel
  Arms: Liposomal bupivacaine

SUMMARY:
The purpose of this study is to establish a relationship between liposomal bupivacaine surgical site injection and postop opioid utilization.

DETAILED DESCRIPTION:
Multiple studies have shown that people who are taking opioids for acute pain have a greater likelihood of long-term opioid use. Many efforts have been made to reduce postop pain and opioid use, including developments in incisional site injections of local anesthetics, continuous incisional site anesthetic pain pumps, as well as multimodal comprehensive pain management, yet patients undergoing lumbar spine surgeries continue to depend on opioids for relief. Liposomal bupivacaine (LB) (Exparel) is a novel formulation of long-acting bupivacaine, lasting for up to 72 hours following injection. LB has been shown to be efficacious in reducing postop pain and opioid utilization in several different surgical settings, however its utility in spine surgeries has still yet to be established. The goal of this study is to determine the efficacy of liposomal bupivacaine vs saline in lumbar spine surgeries in reducing opioid utilization as well as determine if there difference patient reported outcomes and length of hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing isolated lumbar spine procedures using a posterior approach.
* Surgical spine procedures include:
* Single-level lumbar spine surgeries with or without fusion
* Multi-level lumbar spine surgeries with or without fusion

Exclusion Criteria:

* Procedures involving intrathecal space
* Patients with documented allergy to local anesthetics (bupivacaine, lidocaine, procaine, benzocaine).
* Acute lumbar trauma that requires immediate spine stabilization
* Revision of failed back surgeries (including nonunion and malunion)
* Revision of wound or hardware
* Contraindication to regional anesthesia
* Patients with chronic use of opioid medications
* Liver dysfunction (INR > 1.5, albumin <2.8g/dl, bilirubin >2mg/dl)
* Renal dysfunction (eGFR < 60ml/min/1.73m2)
* Severe chronic obstructive pulmonary disease requiring continuous oxygen supplementation
* Unable to give informed consent
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2022-06-13 (Actual); Study Completion 2022-06-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theodore Choma, MD, Principal Investigator — University of Missouri - Missouri Orthopaedic Institute
Locations (1):
- Missouri Orthopaedic Institute, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Butz DR, Shenaq DS, Rundell VL, Kepler B, Liederbach E, Thiel J, Pesce C, Murphy GS, Sisco M, Howard MA. Postoperative Pain and Length of Stay Lowered by Use of Exparel in Immediate, Implant-Based Breast Reconstruction. Plast Reconstr Surg Glob Open. 2015 Jun 5;3(5):e391. doi: 10.1097/GOX.0000000000000355. eCollection 2015 May. PMID 26090281
- [Result] Reynolds RA, Legakis JE, Tweedie J, Chung Y, Ren EJ, Bevier PA, Thomas RL, Thomas ST. Postoperative pain management after spinal fusion surgery: an analysis of the efficacy of continuous infusion of local anesthetics. Global Spine J. 2013 Mar;3(1):7-14. doi: 10.1055/s-0033-1337119. Epub 2013 Mar 2. PMID 24436846
- [Result] Grant GJ, Barenholz Y, Bolotin EM, Bansinath M, Turndorf H, Piskoun B, Davidson EM. A novel liposomal bupivacaine formulation to produce ultralong-acting analgesia. Anesthesiology. 2004 Jul;101(1):133-7. doi: 10.1097/00000542-200407000-00021. PMID 15220782
- [Result] Surdam JW, Licini DJ, Baynes NT, Arce BR. The use of exparel (liposomal bupivacaine) to manage postoperative pain in unilateral total knee arthroplasty patients. J Arthroplasty. 2015 Feb;30(2):325-9. doi: 10.1016/j.arth.2014.09.004. Epub 2014 Sep 16. PMID 25282071
- [Result] American Society of Anesthesiologists Task Force on Acute Pain Management. Practice guidelines for acute pain management in the perioperative setting: an updated report by the American Society of Anesthesiologists Task Force on Acute Pain Management. Anesthesiology. 2012 Feb;116(2):248-73. doi: 10.1097/ALN.0b013e31823c1030. No abstract available. PMID 22227789

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Liposomal Bupivacaine | Placebo Group
Started | 17 | 17
Completed | 17 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Liposomal Bupivacaine | Placebo Group | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 16
  >=65 years | 9 | 9 | 18
Age, Continuous [Mean (Full Range); unit: years] | 63 [38 to 78] | 65 [49 to 76] | 64 [38 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 5 | 5 | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 17 | 17 | 34

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Opioid Utilization
Description: Comparing post operative opioid usage reduction between treatment and placebo group.
Time Frame: Until final follow-up, up to 8 weeks.
Population: Discrepancy comes from patients not reporting morphine milligram equivalents on survey.
Measure: Mean (Standard Deviation); unit: morphine milligram equivalents
Arm/Group | Placebo Group | Liposomal Bupivacaine
Number analyzed (Participants) | 14 | 15
morphine milligram equivalents | 4.82 (10.02) | 9.17 (19.36)

2. Secondary Outcome: Post Operative Pain Scores
Description: Comparing post operative pain scores between treatment and placebo group. Using Visual Analogue Scale (VAS) pain score with scale 0 to 10 with 0 being no pain and 10 being the worst pain of your life.
Time Frame: Until final follow-up or up to 8 weeks after surgery date, whichever comes first.
Population: Reason for participant discrepancy is patients did not fill our VAS pain score survey following surgery.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo Group | Liposomal Bupivacaine
Number analyzed (Participants) | 15 | 16
score on a scale | 4.80 (1.92) | 4.05 (1.74)

3. Secondary Outcome: Length of Stay
Description: Determining how long patient is in hospital.
Time Frame: Until final follow-up, up to 8 weeks.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Placebo Group | Liposomal Bupivacaine
Number analyzed (Participants) | 17 | 17
Hours | 42.69 (40.62) | 29.51 (19.32)

4. Secondary Outcome: Operative Data and Complications
Description: Comparing intraoperative complications, acute postoperative complication, and opioid complications.
Time Frame: Until final follow-up, up to 8 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Group | Liposomal Bupivacaine
Number analyzed (Participants) | 17 | 17
Participants
  Intraoperative Complications: None | 17 | 17
  Intraoperative Complications: Yes | 0 | 0
  Acute Postoperative Complication: None | 15 | 16
  Acute Postoperative Complication: Yes | 2 | 1
  Opioid Complications: None | 17 | 17
  Opioid Complications: Yes | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for a period of 8 weeks.
Description: Our definition of an adverse event did not differ from the definition given by clinicaltrials.gov.
Arm/Group | Liposomal Bupivacaine | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 0/17 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-25): https://cdn.clinicaltrials.gov/large-docs/96/NCT04644796/Prot_SAP_000.pdf